CLINICAL TRIAL: NCT02325622
Title: Relationships Between Mean Plasma Glucose and HbA1c in Compensated and Decompensated Cirrhotic Patients With Hepatogenous Diabetes
Brief Title: Relationships Between Mean Plasma Glucose and HbA1c in Cirrhotic Patients With Hepatogenous Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Moon Young Kim, MD.,PhD, Yonsei University
Other Study IDs: A1C-2014
Record Dates: First submitted 2014-12-16; First posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Liver Cirrhosis; Diabetes Mellitus
MeSH Terms: conditions — Liver Cirrhosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — LSP, fructosamine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The liver plays a crucial role in physiological glycemic control through its involvement in several glucose metabolism processes, including glycogenogenesis and glycogenolysis. Liver diseases result in impaired glucose metabolism due to hepatocyte dysfunction, termed as "hepatogenous diabetes". Abnormal glucose metabolism is found in over 90% of patients with liver cirrhosis. and clinically significant diabetes is known to occur in 30% to 70% of the patients.

A cohort study of cirrhotic patients with hepatogenous diabetes reported a relatively low diabetic complication rate, and the majority of mortality causes were complications related to liver cirrhosis; furthermore, mortality rate due to diabetic complications were reported to be low. Nonetheless, the average survival rate following the diagnosis of liver cirrhosis is rising due to increasing early detection rate and improvements in treatment modalities, and such rise in survival is expected to result in increased prevalence of hepatogenous diabetes and its complications. Therefore, it is necessary to formulate an accurate diagnosis of hepatogenous and to provide appropriate treatment.

Analyses of the Diabetes Control and Complications Trial (DCCT) demonstrated an association between glycated hemoglobin (HbA1c) and mean plasma glucose concentration in diabetic patients, and currently, HbA1c is being employed as an appropriate marker in diagnosing diabetes mellitus and in monitoring the control of mean blood glucose.

The association between mean plasma glucose concentration and HbA1c in cirrhotic patients has not been clearly established as of yet; however, HbA1c in cirrhotic patients is expected to be influenced by various factors resulted by liver cirrhosis and splenomegaly, including rapid erythrocyte turnover rate and other glycation processes.

Therefore, HbA1c may not be an appropriate indicator in the diagnosis of hepatogenous diabetes or the monitoring of glycemic control; however, no systemic study on this issue has been performed so far. Therefore, the investigators are aiming to investigate the association between mean plasma glucose concentration and HbA1c in patients with compensated or decompensated liver cirrhosis who also have hepatogenous diabetes.

DETAILED DESCRIPTION:
1. Primary end outcome Association between mean plasma glucose concentration and glycated hemoglobin in patients with compensated or decompensated liver cirrhosis who also have hepatogenous diabetes
2. Secondary end outcome

   1. HbA1c distribution in patients diagnosed with hepatogenous diabetes confirmed by 75-gram oral glucose tolerance test (OGTT)
   2. Association between mean preprandial blood glucose concentration and glycated hemoglobin in patients with compensated or decompensated liver cirrhosis who also have hepatogenous diabetes
   3. Association between mean postprandial blood glucose concentration and glycated hemoglobin in patients with compensated or decompensated liver cirrhosis who also have hepatogenous diabetes
   4. Association between mean plasma glucose concentration and glycated hemoglobin according to Child-pugh's classification and liver stiffness severity
   5. Factors contributing to discrepancy between mean plasma glucose concentration and HbA1c in patients with compensated or decompensated liver cirrhosis who also have hepatogenous diabetes

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Age greater than 20 years and less than 70 years
* Diabetes mellitus that occurred after the diagnosis of liver cirrhosis
* Diagnostic criteria for diabetes mellitus

  * Fasting plasma glucose ≥ 126 mg/dL
  * 2-hour plasma glucose ≥ 200 mg/dL after 75-g OGTT
* Able to consent to study participation (either by the patient him/herself or by legal guardian)

Exclusion Criteria:

* Patients in shock requiring vasopressors
* Patients with heart or respiratory failure
* Patients with uncontrolled infection (such as spontaneous bacterial peritonitis)
* Patients with acute renal failure due to medication or renal causes
* Hemoglobin ≤ 10mg/dl
* Patients using insulin, steroid, or beta-blockers
* History of hepatocellular carcinoma or other malignancies, or history of diagnosed malignancy that has not been completely remitted
* Patients with medical or psychiatric problems that disables them from performing clinical trial
* Pregnant or lactating women
* Patients unable to comply to trial plan or follow-up monitoring
* Patients deemed by the investigator(s) to be inappropriate for study participation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver cirrhosis diagnosed after combining clinical symptoms (thrombocytopenia, gastric/esophageal varices, ascites), histologic studies, and imaging studies (ultrasound, Fibroscan)
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Association between mean plasma glucose concentration and glycated hemoglobin in cirrhosis | 3 months
  The patient choose 3 days within each month, during which they shall check blood glucose level 7 times daily (fasting and 2-hour postprandial glucose for each meal plus bedtime glucose). This shall be done for 3 months.
  The study shall be concluded after laboratory studies, including glycated hemoglobin, after 3 months.
  Safety assessment :
  The subjects shall be educated on hypoglycemic symptoms, checking blood glucose upon onset of hypoglycemia, and immediate food intake. They shall also be instructed to report such events immediately by phone. The cause of hypoglycemia shall be evaluated, and the medications shall be adjusted.
  Efficacy assessment :
  To assess the primary outcome, the mean plasma glucose shall be calculated by first obtaining the mean of self-monitored blood glucose across 3 days every month and then by adding 11% of the value to the mean- this shall be compared with glycated hemoglobin level measured at 3 months after baseline to check for association.

CONTACTS AND LOCATIONS:
Overall Officials: Moon Young Kim, MD. PhD, Principal Investigator — Department of Internal Medicine, Wonju Severance Christian Hospital
Locations (1):
- Yonsei University Wonju Severance Cristian Hospital, Wŏnju, Gangwon-do, South Korea

REFERENCES:
- [Background] Rohlfing CL, Wiedmeyer HM, Little RR, England JD, Tennill A, Goldstein DE. Defining the relationship between plasma glucose and HbA(1c): analysis of glucose profiles and HbA(1c) in the Diabetes Control and Complications Trial. Diabetes Care. 2002 Feb;25(2):275-8. doi: 10.2337/diacare.25.2.275. PMID 11815495
- [Background] Kilpatrick ES, Rigby AS, Atkin SL. Variability in the relationship between mean plasma glucose and HbA1c: implications for the assessment of glycemic control. Clin Chem. 2007 May;53(5):897-901. doi: 10.1373/clinchem.2006.079756. Epub 2007 Mar 23. PMID 17384010
- [Background] Koga M, Kasayama S, Kanehara H, Bando Y. CLD (chronic liver diseases)-HbA1C as a suitable indicator for estimation of mean plasma glucose in patients with chronic liver diseases. Diabetes Res Clin Pract. 2008 Aug;81(2):258-62. doi: 10.1016/j.diabres.2008.04.012. Epub 2008 Jun 2. PMID 18513821
- [Background] Bando Y, Kanehara H, Toya D, Tanaka N, Kasayama S, Koga M. Association of serum glycated albumin to haemoglobin A1C ratio with hepatic function tests in patients with chronic liver disease. Ann Clin Biochem. 2009 Sep;46(Pt 5):368-72. doi: 10.1258/acb.2009.008231. Epub 2009 Aug 12. PMID 19675058
- [Background] Lahousen T, Hegenbarth K, Ille R, Lipp RW, Krause R, Little RR, Schnedl WJ. Determination of glycated hemoglobin in patients with advanced liver disease. World J Gastroenterol. 2004 Aug 1;10(15):2284-6. doi: 10.3748/wjg.v10.i15.2284. PMID 15259084